CLINICAL TRIAL: NCT00221260
Title: Perioperative Epidural Trial (POET) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Dr. Peter Choi, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C04-0078; 04-3046
Record Dates: First submitted 2005-09-18; First posted 2005-09-22 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Post Operative Pain Control
Keywords: Analgesia; anesthesia
MeSH Terms: conditions — Agnosia | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: anesthesia — Intraoperative general anesthesia AND postoperative IV narcotic analgesia.

SUMMARY:
To investigate if the use of perioperative neuraxial blockade reduces post-operative mortality and cardiorespiratory events compared to intraoperative general anesthesia AND postoperative IV narcotic analgesia. This is a feasibility study to determine if recruitment and execution of the protocol could be done in a timely manner in a much larger trial

ELIGIBILITY:
Inclusion Criteria:

Subjects at high risk of cardio-respiratory complications post operatively.

Exclusion Criteria:

Contraindication to epidural anesthesia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Combined mortality, MI, cardiac arrest, post operative pneumonia , and respiratory failure

SECONDARY OUTCOMES:
DVT, pulmonary embolism, TIA, CVA, CHF, clinically significant bradycardia/hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Peter Choi, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Clinical Health Research Unit, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Choi PT, Beattie WS, Bryson GL, Paul JE, Yang H. Effects of neuraxial blockade may be difficult to study using large randomized controlled trials: the PeriOperative Epidural Trial (POET) Pilot Study. PLoS One. 2009;4(2):e4644. doi: 10.1371/journal.pone.0004644. Epub 2009 Feb 27. PMID 19247497